CLINICAL TRIAL: NCT03767309
Title: Management of Miller Class I & II Gingival Recession Using Conventional Versus Abrasive De-epithelization of Palatal Graft
Brief Title: Management of Miller Class I & II Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halla Gamal Mohammed Esmail (Other)
Responsible Party: Sponsor-Investigator, Halla Gamal Mohammed Esmail, Dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1788
Record Dates: First submitted 2018-11-29; First posted 2018-12-06 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2018-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): SCTG will be harvested from the palate in the intervention group (coronally advanced flap and abrasively de-epithelialized free gingival graft)
  Interventions: Procedure: coronally advanced flap with abrasive de-epithelized graft.
- Control group (Active Comparator): SCTG will be harvested from the palate using Zucchilli's technique (zucchelli, 2010) in the control group (coronally advanced flap and conventionally de-epithelialized free gingival graft)
  Interventions: Procedure: coronally advanced flap with de-epithelized graft.

INTERVENTIONS:
Procedure: coronally advanced flap with abrasive de-epithelized graft. — SCTG will be harvested from the palate by abrasive de-epithelialization of palatal graft involves removing the epithelium of the selected area with a high-speed hand piece and diamond bur
  Arms: Test group
Procedure: coronally advanced flap with de-epithelized graft. — SCTG will be harvested from the palate by abrasive de-epithelialization of palatal graft involves removing the epithelium of the selected area with a blade
  Arms: Control group

SUMMARY:
Management of Miller class I & II gingival recession using coronally advanced flap combined with conventional de-epithelialized free gingival graft versus coronally advanced flap combined with abrasive de-epithelized connective tissue graft Null hypothesis: In patients with Miller class I and II gingival recession, there is no difference between coronally advanced flap with conventional de-epithelialized free gingival graft and coronally advanced flap with abrasive de-epithelized connective tissue graft in recession depth reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Systemically healthy patients.
* Miller's Class I and II recession defects with recession depth ≥ 2mm.
* Presence of identifiable cemento-enamel junction (CEJ).
* Clinical indication and/or patient request for recession coverage.
* Smoking ≤ 10 cigarettes/day.
* Cooperative patients able and accept to come for follow up appointments.

Exclusion Criteria:

* Pregnant females.
* Smoking ˃ 10 cigarettes/day.
* Contraindication for periodontal surgery.
* Patients with poor oral hygiene.
* Recession defects associated with caries or restoration as well as
* Teeth with evidence of a pulpal pathology
* Molar teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Direct Post-operative pain | 7 days
  Directly will be evaluated post-surgically with Visual Analogue Scale with numbers from 0 to 10 that given to the patients at 7 days follow-up visits.
Indirect Post-operative pain | 7 days
  Indirectly will be evaluated on the basis of the mean consumption of analgesics

SECONDARY OUTCOMES:
Complete Root Coverage | 6 months
  CRC evaluated in patients by single operator clinically using a periodontal probe. Root coverage was deemed complete when the gingival margin is at or above the level of CEJ
Recession depth. | 6 months
  Measured from the CEJ to the most apical extension of the gingival margin
Gingival Recession Width | 6 months
  measured at the level of the CEJ.
Width Of Keratinized Gingiva | 6 months
  Measured from the gingival margin to the mucogingival line
Root Coverage Esthetic Score | 6 months
  The RES system evaluates five variables 6 months following surgery
Gingival thickness | 6 months
  It will be measured by penetrating the gingiva mid-buccally in the attached gingiva, half way between mucogingival junction and free gingival groove with the periodontal probe after giving local anesthesia to measure the thickness of gingival tissues.
Surgical chair time | at the time of surgery
  measured by Stop watch

IPD SHARING:
Plan to Share IPD: Undecided